CLINICAL TRIAL: NCT02124759
Title: Mechanism of Microbiome-induced Insulin Resistance in Humans (Aim 1)
Acronym: MicroB1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20130459H; IRB #20130458H (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Sevelamer; Synbiotics; maltodextrin; Diet, High-Fat; Diet, Fat-Restricted; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo: maltodextrin, 6 g three times a day
  Interventions: Drug: Maltodextrin; Other: High Fat diet; Other: Low Fat diet
- Sevelamer (Active Comparator): Sevelamer: (1.6 g sevelamer + 4.4 g maltodextrin three times a day)
  Interventions: Drug: Sevelamer; Other: High Fat diet; Other: Low Fat diet
- Synbiotic (Active Comparator): Synbiotic: 5g Oligofructose + 4x1010 Bifidobacterium longum CFU 3x daily during diet
  Interventions: Drug: Synbiotic; Other: High Fat diet; Other: Low Fat diet

INTERVENTIONS:
Drug: Sevelamer — 1.6 g sevelamer + 4.4 g maltodextrin three times a day
  Other Names: Renvela
  Arms: Sevelamer
Drug: Synbiotic — 5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming units (CFU)/g) three times a day.
  Arms: Synbiotic
Drug: Maltodextrin — This is a control group. Maltodextrin, 6 g three times a day
  Arms: Placebo
Other: High Fat diet — The High Fat diet consists of 60% energy from fat (50% saturated), 15% of energy as carbohydrate and 25% from protein consumed while study intervention is being administered.
  Other Names: Isocaloric high fat diet
Other: Low Fat diet — The isocaloric low fat diet will provide 55% energy from carbohydrates, 20% from fat and 25% from protein.
  Other Names: Isocaloric low fat (normal) diet

SUMMARY:
The purpose of this study is to determine insulin sensitivity in individuals that are lean normal glucose tolerant subjects after consumption of a normal low fat diet and after a high fat diet and to explore the effects of high fat consumption on the intestinal microbiome, and metabolic endotoxemia.( Aim 1 of the protocol, a separate record is available for Aim 2)

DETAILED DESCRIPTION:
We will test the hypothesis that a high fat diet given to lean, normal glucose tolerant subjects will impair insulin signaling and sensitivity and modify gut microbiome composition and enhance intestinal permeability, which will increase plasma LPS concentration, induce an inflammatory response in peripheral tissues (skeletal muscle). Also we will test the hypothesis that the inflammatory response and insulin resistance caused by high fat ingestion can be ameliorated by administering

* a synbiotic (Bifidobacterium longum R0175 and oligofructose) which protects the intestinal epithelial barrier and decreases intestinal translocation of LPS; and
* sevelamer, an agent which sequesters lipopolysaccharide (LPS) in the gastrointestinal tract limiting its translocation into the circulation.

All subjects are fed both a low fat diet (considered a normal diet) and high fat diet, first one and then the other in no particular sequence. After a washout period participants are fed the other type of high or low fat diet, depending on which diet they were first assigned to in order to compare the effects of the intervention on insulin sensitivity during each diet.

ELIGIBILITY:
Inclusion Criteria:

* Both genders. All races and ethnic groups.
* Premenopausal women in the follicular phase, non-lactating, and with a negative pregnancy test. Postmenopausal women on stable dose of or not exposed to hormone replacement for ≥6 months.
* Hematocrit (HCT)≥ 34%, serum creatinine ≤ 1.4 mg/dl, and normal serum electrolytes, urinalysis, and coagulation tests. Liver function tests (LFTs) up to 2 times normal.
* Stable body weight (±2%) for ≥ 3 months
* Two or less sessions of strenuous exercise/wk for last 6 months.

Exclusion Criteria:

* Presence of diabetes or impaired glucose tolerance based on ADA criteria.
* Current treatment with drugs known to affect glucose and lipid homeostasis. If the subject has been on a stable dose for the past 3 months, the following agents will be permitted: calcium channel blockers, β-blockers, ACE inhibitors, angiotensin receptor blockers, and statins
* History of allergy to sevelamer.
* History of Non-steroidal anti-inflammatory drugs or systemic steroid use for more than a week within 3 months.
* Current treatment with anticoagulants (warfarin). Aspirin (up to 325 mg) and clopidogrel will be permitted if these can be held for seven days prior to the biopsy in accordance with the primary physician.
* Use of agents that affect gut flora (e.g. antibiotics, colestyramine, lactulose, PEG) within 3 months.
* History of heart disease (New York Heart Classification greater than grade II; more than non-specific ST-T wave changes on the ECG), peripheral vascular disease, pulmonary disease, smokers.
* Poorly controlled blood pressure (systolic BP>170, diastolic BP>95 mmHg).
* Active inflammatory, autoimmune, hepatic, gastrointestinal, malignant, and psychiatric disease.
* History of gastrointestinal surgery or gastrointestinal obstruction within two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Audie L. Murphy VA Hospital, STVHCS, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were initially screened by BMI and glucose tolerance via OGTT. Qualified Study participants were then assigned to begin a low or high isocaloric diet and then randomized to one of the 3 arms for 4 weeks. After a 10-12 week washout, subjects are changed over to the other diet and remain in the same arm of the study that they were in previously.
Groups:
- Placebo: placebo, maltodextrin, 6 g three times a day during diet
  This is a control group.
- Sevelamer: Sevelamer: 1.6 g sevelamer + 4.4 g maltodextrin three times a day during diet
- Synbiotic: 5g Oligofructose + 4x1010 Bifidobacterium longum CFU 3x daily during diet
Period: Overall Study
Arm/Group | Placebo | Sevelamer | Synbiotic
Started (Subjects gave informed consent to be screened for study.) | 6 | 7 | 7
Subjects Randomized to Intervention | 4 | 5 | 4
Low Fat Diet | 4 (2 subjects did not complete and were withdrawn) | 4 | 4
High Fat Diet | 2 (1 subject did not complete) | 5 (One subject withdrew (low fat diet had already been completed)) | 4 (One subject withdrew and did not complete the low fat diet)
Completed | 1 | 4 | 3
Not Completed | 5 | 3 | 4
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Screen Fail | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline participants were consented and passed screening and completed both high fat and low fat diet while randomized to one of the interventions.
Groups:
- Placebo: placebo, maltodextrin, 6 g three times a day
- Synbiotic: *synbiotic [5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion CFU/g)three times a day]
- Total: Total of all reporting groups
Arm/Group | Placebo | Sevelamer | Synbiotic | Total
Number analyzed (Participants) | 1 | 4 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (0) | 40.5 (22.0) | 59 (3.8) | 50.6 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 7
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 4
  Not Hispanic or Latino | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 5
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Low Fat Diet
Description: Skeletal muscle insulin sensitivity measured after 28 days of low fat diet and drug intervention. The isocaloric low fat diet will provide 55% energy from carbohydrates, 20% from fat and 25% from protein.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: M value (mg/kg/min
Arm/Group | Placebo | Sevelamer | Synbiotic
Number analyzed (Participants) | 1 | 4 | 3
M value (mg/kg/min | 6.5 (0) | 8.2 (2.4) | 9.8 (0.6)

2. Primary Outcome: Insulin Sensitivity High Fat Diet
Description: Skeletal muscle insulin sensitivity measured after 28 days of high fat diet. The High Fat diet consists of 60% energy from fat (50% saturated), 15% of energy as carbohydrate and 25% from protein consumed while study intervention is being administered.
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: M Value (mg/kg/min)
Arm/Group | Placebo | Sevelamer | Synbiotic
Number analyzed (Participants) | 1 | 4 | 3
M Value (mg/kg/min) | 6.8 (0) | 8.5 (1.87) | 8.8 (1.63)
Statistical Analysis 1: Comparison: Placebo vs Sevelamer vs Synbiotic; Null hypothesis is that high fat diet will have no effect on M value, the measure of insulin sensitivity for each intervention as assessed by clamp; Test type: Superiority; p > 0.05, t-test, 2 sided; Paired T-test

3. Secondary Outcome: Plasma Endotoxin Levels
Description: Endotoxin is a bacterially derived product that we hypothesized would impact insulin sensitivity through pro inflammatory pathways.
Time Frame: At baseline, on day 3, and 28 of the intervention.
Population: Plasma Endotoxin levels not analyzed after study completed enrollment due to low subject enrollment and limited ability to compare between subjects (max n=3 per group)
Groups:
- Placebo: The high fat diet will provide 60% of energy from fat (of which 50% from saturated fat), 15% of energy as CHO and 25% from protein.
  subjects will be randomized to receive, in a double-blind fashion
  Maltodextrin: This is a control group. Maltodextrin, 6 g three times a day
- Sevelamer: The high fat diet will provide 60% of energy from fat (of which 50% from saturated fat), 15% of energy as CHO and 25% from protein.
  subjects will be randomized to receive, in a double-blind fashion Sevelamer: 1.6 g sevelamer + 4.4 g maltodextrin three times a day
- Synbiotic: The high fat diet will provide 60% of energy from fat (of which 50% from saturated fat), 15% of energy as CHO and 25% from protein.
  subjects will be randomized to receive, in a double-blind fashion Synbiotic: 5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming units (CFU)/g) three times a day.
Arm/Group | Placebo | Sevelamer | Synbiotic
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Gut Permeability
Description: Gut permeability is measured using a lactulose/mannitol ingestion assay where urine samples are collected to analyse the ratio of excreted lactulose:mannitol.
Time Frame: on Day 24 of the intervention.
Population: Gut permeability not analyzed after study completed enrollment due to low subject enrollment and limited ability to compare between subjects (max n=3 per group)
Arm/Group | Placebo | Sevelamer | Synbiotic
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected over the course of the study intervention period, beginning with subject's enrollment into study and ending once they completed all visits. This period takes approximately 6 months from screening to completion of all visits.
Description: Adverse events were collected per arm of the study, for placebo, sevelamer and synbiotic, rather than by arm and low or high fat diet. Each arm reports adverse events to include the participant assignment to either low or high fat diets.
Groups:
- Placebo: Maltodextrin: This is a control group that were fed both low and high fat diets.
  Maltodextrin, 6 g three times a day
- Sevelamer: Sevelamer: 1.6 g sevelamer + 4.4 g maltodextrin three times a day that were fed either a low fat or high fat diet, followed by the other type of diet.
- Synbiotic: Synbiotic: 5 g of oligofructose + 1 g Bifidobacterium longum R0175 (4 billion colony forming units (CFU)/g) three times a day that were fed either a low fat or high fat diet, followed by the other type of diet.
Arm/Group | Placebo | Sevelamer | Synbiotic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/6 | 3/7 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Sevelamer (N=7) | Synbiotic (N=7)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Hematoma at muscle biopsy site
Mouth Ulcers (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ear Itching (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Bloating/Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vasovagal Syncope (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) — Syncope during medical procedure
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gum Infection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Treated with Abx and removed off protocol

LIMITATIONS AND CAVEATS:
Despite continued recruitment efforts, we had difficulty with subjects fully completing the study due to dissatisfaction with the diets. Evaluable subjects completed both low and high fat diet while randomized to one of the three interventions, and only insulin sensitivity was captured for both the low fat and high fat diets due to the low completion numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT02124759/Prot_SAP_000.pdf